CLINICAL TRIAL: NCT02024074
Title: Performance of Tc99m Sestamibi Molecular Breast Imaging (Tc-MBI) Versus Magnetic Resonance Imaging in the Diagnosis of Breast Carcinoma: A Pilot Study
Brief Title: Evaluation of Magnetic Resonance Imaging (MRI) vs Molecular Breast Imaging (Tc-MBI) in Breast Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by the Sponsor due to slow enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Raghuveer Halkar, MD, Professor, School of Medicine, Department of Radiology, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00064317
Record Dates: First submitted 2013-12-23; First posted 2013-12-31 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sestamibi(Tc- MBI) scan of the breast (Other)
  Interventions: Other: Sestamibi (Tc-MBI) scan of the breast

INTERVENTIONS:
Other: Sestamibi (Tc-MBI) scan of the breast — Patients will be given 8mCi of Sestamibi intravenously. following which Sestamibi scan will be performed on the breast. Sestamibi scan will be done prior to any surgical procedure..

SUMMARY:
The objective of this study is to evaluate the usefulness of Tc-99m Sestamibi Molecular Breast Imaging as an imaging modality for breast cancer screening.

Tc-MBI has shown significantly higher sensitivity and equivalent specificity in the detection of breast cancer among high risk women when compared to mammography. However, there is little published data comparing Tc-MBI to MRI for evaluating extent of disease in women with known breast cancer.

The study will target twenty (20) women with newly diagnosed breast cancer who are scheduled to undergo biopsy of additional suspicious lesions that were identified on standard of care contrast- enhanced breast MRI. Prior to the biopsy, these subjects will receive a Tc-MBI scan of the breast. The results from both imaging methods will be compared to histological findings. These results may be used to design larger and more comprehensive studies with an overarching goal to determine if there is a role for Tc-MBI in the pre-operative evaluation of patients with known breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Women Patients must be 18 years of age or older. Patients will have biopsy proven unilateral breast cancer with ipsilateral or contralateral suspicious lesions on contrast-enhanced breast MRI and be a candidate for additional tissue biopsy.

Patients must be able to remain still for Tc-MBI scanning Patients must be able to provide written informed consent

Exclusion Criteria:

Men, age less than 18, inability to remain still for Tc-MBI scanning, cannot provide written informed consent, known untreated bilateral breast cancer, evidence of distant metastasis disease (M=1), pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cancer detection rates by Sestambi imaging | Up to 2 years
  This study will determine whether Tc-MBI is useful in the pre-operative evaluation of patients with known breast cancer. Patients will be tracked for 2 years to see if histological evidence is found to confirm Tc-MBI findings

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States